CLINICAL TRIAL: NCT01844856
Title: A Phase 3, Randomized, Double-Blind, Double-Dummy, Multicenter, Prospective Study to Assess the Efficacy and Safety of Eravacycline Compared With Ertapenem in Complicated Intra-abdominal Infections
Brief Title: Efficacy and Safety Study of Eravacycline Compared With Ertapenem in Complicated Intra-abdominal Infections
Acronym: IGNITE1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Organization: La Jolla Pharmaceutical Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP-434-008
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Complicated Intra-abdominal Infections
MeSH Terms: interventions — eravacycline; Ertapenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eravacycline, 1.0 mg/kg q12h (Experimental): Eravacycline was administered intravenously (IV) at a dose of 1.0 milligram per kilogram of body weight (mg/kg) every 12 hours (q12h) for a minimum of 4 days and a maximum of 14 days. Eravacycline treatment was to be stopped when symptoms of complicated intra-abdominal infection (cIAI) resolved, there was treatment failure, or the maximum allowed number of infusion days was reached.
  Interventions: Drug: Eravacycline; Drug: Placebo
- Ertapenem, 1.0 g q24h (Active Comparator): Ertapenem was administered IV at a dose of 1.0 gram (g) every 24 hours (q24h) for a minimum of 4 days and a maximum of 14 days. Ertapenem treatment was to be stopped when symptoms of cIAI resolved, there was treatment failure, or the maximum allowed number of infusion days was reached.
  Interventions: Drug: Ertapenem; Drug: Placebo

INTERVENTIONS:
Drug: Eravacycline
  Other Names: TP-434
  Arms: Eravacycline, 1.0 mg/kg q12h
Drug: Ertapenem
  Other Names: Invanz
  Arms: Ertapenem, 1.0 g q24h
Drug: Placebo — Administered IV to maintain the blind.

SUMMARY:
This is a Phase 3, randomized, double-blind, double-dummy, multicenter, prospective study to assess the efficacy, safety, and pharmacokinetics of eravacycline compared with ertapenem in the treatment of adult complicated intra-abdominal infections (cIAI).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant hospitalized for cIAI
2. At least 18 years of age (and not over 65 years of age for participant in India)
3. Evidence of a systemic inflammatory response
4. Abdominal pain or flank pain (with or without rebound tenderness), or pain caused by cIAI that is referred to another anatomic area
5. Able to provide informed consent
6. If male: must agree to use an effective barrier method of contraception during the study and for 90 days following the last dose if sexually active with a female of childbearing potential
7. If female, not pregnant or nursing or, if of childbearing potential: either will commit to use at least two medically accepted, effective methods of birth control (for example, condom, oral contraceptive, indwelling intrauterine device, hormonal implant /patch, injections, approved cervical ring) during study drug dosing and for 90 days following last study drug dose or practicing sexual abstinence

Exclusion Criteria:

1. Unlikely to survive the 6-8 week study period
2. Renal failure
3. Presence or possible signs of hepatic disease
4. Immunocompromised condition, including known human immunodeficiency virus (HIV) positivity (requiring anti-retroviral therapy or with CD4 count <300), acquired immune deficiency syndrome (AIDS), organ (bone marrow) transplant recipients, and hematological malignancy. Immunosuppressive therapy, including use of high-dose corticosteroids (for example, >40 mg prednisone or equivalent per day for greater than 2 weeks)
5. History of hypersensitivity reactions to tetracyclines, carbapenems, β-lactam antibiotics or to excipients contained in the study drug formulations
6. Participation in any investigational drug or device study within 30 days prior to study entry
7. Known or suspected current Central Nervous System disorder that may predispose to seizures or lower seizure threshold
8. Previously received eravacycline in a clinical trial
9. Antibiotic-related exclusions:

   1. Receipt of effective antibacterial drug therapy for cIAI for a continuous duration of >24 hours during the 72-hour preceding enrollment (however, participants with documented cIAI [that is, known baseline pathogen] who have received at least 72 hours of antibiotic therapy and are considered treatment failures may be enrolled. Treatment failure is defined as persistent fever and/or clinical symptoms; or the development of a new intra-abdominal abscess after ≥72 hours of antibiotic therapy), or
   2. Receipt of ertapenem or any other carbapenem, or tigecycline for the current infection or
   3. Need for concomitant systemic antimicrobial agents other than study drug
10. Refusal of mechanical ventilation, dialysis or hemofiltration, cardioversion or any other resuscitative measures and drug/fluid therapy at time of consent
11. Known or suspected inflammatory bowel disease or associated visceral abscess
12. The anticipated need for systemic antibiotics for a duration of more than 14 days
13. Systemic malignancy that required chemotherapy, immunotherapy, radiation therapy or antineoplastic therapy within the previous 3 months or that is anticipated to begin prior to the Test-of-Cure (TOC) visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick T Horn, MD, PhD, Study Director — Tetraphase Pharmaceuticals, Inc
Locations (69):
- United States (19):
  - Florence, Alabama
  - Mobile, Alabama
  - Glendale, California
  - La Mesa, California
  - Los Angeles, California
  - Torrance, California
  - Aurora, Illinois
  - Carmel, Indiana
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Minneapolis, Minnesota
  - Las Vegas, Nevada
  - Camden, New Jersey
  - Teaneck, New Jersey
  - Cleveland, Ohio
  - Columbus, Ohio
  - Weston, Ohio
  - Houston, Texas
  - Seattle, Washington
- Córdoba, Argentina
- Bulgaria (5):
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Varna
- Czechia (6):
  - Brno
  - Kladno
  - Mělník
  - Olomouc
  - Prague
  - Ústí nad Labem
- Estonia (3):
  - Kohtla-Järve
  - Tallinn
  - Tartu
- Paris, France
- Germany (3):
  - Heidelberg
  - Lübeck
  - Magdeburg
- Latvia (3):
  - Daugavpils
  - Liepāja
  - Riga
- Lithuania (4):
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Vilnius
- Romania (4):
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Timișoara
- Russia (9):
  - Kaluga
  - Kemerovo
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Smolensk
  - Tomsk
  - Volgograd
  - Vsevolozhsk
- South Africa (4):
  - Benoni
  - Johannesburg
  - Pretoria
  - Worcester
- Ukraine (7):
  - Dnipropetrovsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Odesa
  - Uzhhorod
  - Zaporizhia

REFERENCES:
- [Derived] Solomkin JS, Sway A, Lawrence K, Olesky M, Izmailyan S, Tsai L. Eravacycline: a new treatment option for complicated intra-abdominal infections in the age of multidrug resistance. Future Microbiol. 2019 Oct;14:1293-1308. doi: 10.2217/fmb-2019-0135. Epub 2019 Oct 1. PMID 31570004
- [Derived] Solomkin JS, Gardovskis J, Lawrence K, Montravers P, Sway A, Evans D, Tsai L. IGNITE4: Results of a Phase 3, Randomized, Multicenter, Prospective Trial of Eravacycline vs Meropenem in the Treatment of Complicated Intraabdominal Infections. Clin Infect Dis. 2019 Aug 30;69(6):921-929. doi: 10.1093/cid/ciy1029. PMID 30561562
- [Derived] Solomkin J, Evans D, Slepavicius A, Lee P, Marsh A, Tsai L, Sutcliffe JA, Horn P. Assessing the Efficacy and Safety of Eravacycline vs Ertapenem in Complicated Intra-abdominal Infections in the Investigating Gram-Negative Infections Treated With Eravacycline (IGNITE 1) Trial: A Randomized Clinical Trial. JAMA Surg. 2017 Mar 1;152(3):224-232. doi: 10.1001/jamasurg.2016.4237. PMID 27851857

RESULTS

PARTICIPANT FLOW:
Groups:
- Eravacycline, 1.0 mg/kg q12h: Eravacycline was administered intravenously (IV) at a dose of 1.0 milligrams per kilogram of body weight (mg/kg) every 12 hours (q12h) for a minimum of 4 days and a maximum of 14 days.
- Ertapenem, 1.0 g q24h: Ertapenem was administered IV at a dose of 1.0 grams (g) every 24 hours (q24h) for a minimum of 4 days and a maximum of 14 days.
Period: Overall Study
Arm/Group | Eravacycline, 1.0 mg/kg q12h | Ertapenem, 1.0 g q24h
Started | 270 | 271
Received at Least 1 Dose of Study Drug | 270 | 268
Completed | 246 | 255
Not Completed | 24 | 16
Not completed — Lost to Follow-up | 15 | 3
Not completed — Adverse Event | 3 | 6
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Noncompliance | 2 | 3
Not completed — Enterococcus Resistant | 0 | 1
Not completed — Inadvertently Not Scheduled | 1 | 0
Not completed — Randomized but was a Screen Failure | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants (Intent-to-treat [ITT] population)
Groups:
- Eravacycline, 1.0 mg/kg q12h: Eravacycline was administered IV at a dose of 1.0 mg/kg q12h for a minimum of 4 days and a maximum of 14 days.
- Ertapenem, 1.0 g q24h: Ertapenem was administered IV at a dose of 1.0 g q24h for a minimum of 4 days and a maximum of 14 days.
- Total: Total of all reporting groups
Arm/Group | Eravacycline, 1.0 mg/kg q12h | Ertapenem, 1.0 g q24h | Total
Number analyzed (Participants) | 270 | 271 | 541
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean/standard deviation of age for the combined eravacycline and ertapenem treatment groups was calculated by hand.
  years | 54.8 (16.92) | 54.8 (16.09) | 54.8 (16.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 108 | 222
  Male | 156 | 163 | 319
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 261 | 262 | 523
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 263 | 260 | 523
  Black or African American | 1 | 3 | 4
  Asian | 1 | 3 | 4
  Other Race | 4 | 5 | 9
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Russian Federation | 28 | 24 | 52
  Romania | 42 | 42 | 84
  United States | 18 | 20 | 38
  Ukraine | 38 | 38 | 76
  Czech Republic | 14 | 17 | 31
  Latvia | 25 | 23 | 48
  South Africa | 0 | 1 | 1
  Bulgaria | 45 | 44 | 89
  Lithuania | 26 | 26 | 52
  Germany | 2 | 2 | 4
  Estonia | 32 | 34 | 66

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response of Eravacycline and Ertapenem Treatment Arms at the Test-of-cure (TOC) Visit in the Microbiological Intent-to-treat (Micro-ITT) Population
Description: Clinical response was classified as cure (complete resolution or significant improvement of signs and symptoms of the index infection), failure (death related to complicated intra-abdominal infection [cIAI], unplanned surgical procedures or percutaneous drainage procedures, persisting or recurrent infection within the abdomen, postsurgical wound infection, or administration of effective concomitant antibacterial therapy), or indeterminate (outcome was neither cure nor failure, or assessment was not available). Participants who were failures at the End-of-Treatment (EOT) visit (within 24 hours of last dose) were considered failures at the TOC visit. The number of participants with a clinical response classification of cure, failure, or indeterminate is presented.
Time Frame: TOC visit: 25-31 days after the first dose of study drug
Population: All randomized participants who had baseline bacterial pathogens that cause cIAI and against at least one of which the investigational drug has in vitro antibacterial activity (micro-ITT population).
Measure: Number; unit: participants
Arm/Group | Eravacycline, 1.0 mg/kg q12h | Ertapenem, 1.0 g q24h
Number analyzed (Participants) | 220 | 226
participants
  Cure | 191 | 198
  Failure | 19 | 11
  Indeterminate | 10 | 17

2. Secondary Outcome: Clinical Response of Eravacycline and Ertapenem Treatment Arms in the Modified Intent-to-treat (MITT) Population at the TOC Visit
Description: Clinical response was classified as cure (complete resolution or significant improvement of signs and symptoms of the index infection), failure (death related to complicated intra-abdominal infection [cIAI], unplanned surgical procedures or percutaneous drainage procedures, persisting or recurrent infection within the abdomen, postsurgical wound infection, or administration of effective concomitant antibacterial therapy), or indeterminate (outcome was neither cure nor failure, or assessment was not available). Participants who were failures at the EOT visit (within 24 hours of last dose) were considered failures at the TOC visit. The number of participants with a clinical response classification of cure, failure, or indeterminate is presented.
Time Frame: TOC visit: 25-31 days after first dose
Population: All randomized participants who received at least 1 dose of study drug (MITT population).
Measure: Number; unit: participants
Arm/Group | Eravacycline, 1.0 mg/kg q12h | Ertapenem, 1.0 g q24h
Number analyzed (Participants) | 270 | 268
participants
  Cure | 235 | 238
  Failure | 19 | 15
  Indeterminate | 16 | 15

3. Secondary Outcome: Clinical Response of Eravacycline and Ertapenem Treatment Arms in the Clinically Evaluable (CE) Population at the TOC Visit
Description: as for outcome 2
Time Frame: TOC visit: 25-31 days after first dose
Population: All randomized participants who had no major protocol deviations (CE population).
Measure: Number; unit: participants
Arm/Group | Eravacycline, 1.0 mg/kg q12h | Ertapenem, 1.0 g q24h
Number analyzed (Participants) | 239 | 238
participants
  Cure | 222 | 225
  Failure | 17 | 13
  Indeterminate | 0 | 0

ADVERSE EVENTS:
Arm/Group | Eravacycline, 1.0 mg/kg q12h | Ertapenem, 1.0 g q24h
Serious Adverse Events (participants affected / at risk) | 17/270 | 16/268
Other Adverse Events (participants affected / at risk) | 43/270 | 28/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eravacycline, 1.0 mg/kg q12h (N=270) | Ertapenem, 1.0 g q24h (N=268)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 0
Oesophageal fistula (Gastrointestinal disorders) | 1 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 2
Empyema (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 1
Peritoneal abscess (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Biliary drainage (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eravacycline, 1.0 mg/kg q12h (N=270) | Ertapenem, 1.0 g q24h (N=268)
Nausea (Gastrointestinal disorders) | 22 | 2
Vomiting (Gastrointestinal disorders) | 11 | 9
Anaemia (Blood and lymphatic system disorders) | 7 | 9
Pyrexia (General disorders) | 6 | 8
Phlebitis (Vascular disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 60 days prior to submitting or presenting a manuscript, poster, presentation, abstract or other materials relating to the Trial, the PI shall provide to Sponsor all such manuscripts and materials, and Sponsor shall have 60 days to review and comment. If requested, the PI shall remove confidential information prior to submitting or presenting the materials, and shall delay publication or presentation for up to 90 days to allow Sponsor to protect its interests in any such materials.